CLINICAL TRIAL: NCT03877562
Title: A Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of CORT118335 on Olanzapine-Induced Weight Gain in Healthy Subjects
Brief Title: The Effect of CORT118335 on Olanzapine-Induced Weight Gain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CORT118335-852; 2019-000633-39 (EudraCT Number)
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Antipsychotic-induced Weight Gain
MeSH Terms: interventions — Olanzapine; CORT118335

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olanzapine plus CORT118335 (Experimental): Participants will receive olanzapine 10 mg oral tablets and double-blind CORT118335 600 mg after breakfast once daily for 14 days.
  Interventions: Drug: Olanzapine; Drug: CORT118335
- Olanzapine plus Placebo (Placebo Comparator): Participants will receive olanzapine 10 mg oral tablets and double-blind placebo matching CORT118335 oral tablets after breakfast once daily for 14 days.
  Interventions: Drug: Olanzapine; Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 10 mg oral tablet
Drug: CORT118335 — CORT118335 600 mg oral tablets administered as 2 X 300 mg or 6 X 100 mg tablets
  Arms: Olanzapine plus CORT118335
Drug: Placebo — Placebo matching CORT118335, 2 or 6 oral tablets, depending on the CORT118335 tablet strength available
  Arms: Olanzapine plus Placebo

SUMMARY:
This study will investigate if there is any difference in the amount of weight gained by participants taking olanzapine with CORT118335 compared with olanzapine with placebo (a dummy test medicine which looks like CORT118335 but contains no active medicine). Safety and tolerability of CORT118335 when taken with olanzapine will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0 to 25.0 kg/m^2, inclusive
* Stable body weight as indicated by assessment at screening and pre-dose
* Able to swallow the size and number of tablets required
* Provide written informed consent and agree to adhere to study restrictions and contraception requirements.

Exclusion Criteria:

* Have received any investigational medicine in a clinical research study within the previous 3 months, or CORT118335 at any time
* Employee, or immediate family member of a study site or Sponsor employee
* Have a pregnant partner
* History of abuse of any drug or alcohol, or regularly consume more than 21 units alcohol/week
* Smokers or users of e-cigarettes and nicotine replacement products within the last 6 months
* Clinically significant abnormal results of clinical laboratory safety tests, electrocardiogram, or measurement of heart rate and blood pressure
* History of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, respiratory, or gastrointestinal disease, neurological or psychiatric disorder
* History of jaundice or gallstones or had a cholecystectomy
* Family history or known risk for narrow angle glaucoma
* Consumed liquorice or other glycyrrhetic acid derivatives regularly in the past 6 months
* Any condition that could be aggravated by glucocorticoid and/or mineralocorticoid antagonism (e.g., asthma, any chronic inflammatory condition, postural hypotension/orthostatic symptoms)
* Presence or history of clinically significant allergy
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Are taking, or have taken, any prescribed or over-the-counter drug within 14 days other than paracetamol or standard dose multivitamins. Longer restrictions apply for some medicines.
* Lactose intolerance.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Body Weight | Pre-dose on Day 1 (Baseline) and Day 15

SECONDARY OUTCOMES:
Percentage of Participants with One or More Adverse Events | Up to Day 28
Percentage of Participants with One or More Serious Adverse Events | Up to Day 28
Percentage of Participants Discontinued from the Study due to an Adverse Event | Up to Day 28
Mean Change from Baseline in Glucose | Pre-dose on Day 1 (Baseline), pre-dose on Days 8, 15, and 28
Mean Change from Baseline in Insulin | Pre-dose on Day 1 (Baseline), pre-dose on Days 8, 15, and 28
Mean Change from Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Pre-dose on Day 1 (Baseline), pre-dose on Days 8, 15, and 28
Mean Change from Baseline in Triglycerides | Pre-dose on Day 1 (Baseline), pre-dose on Days 8, 15, and 28
Mean Change from Baseline in Waist-to-Hip Ratio | Pre-dose on Day 1 (Baseline), Days 8, 15, and 28
Plasma Pharmacokinetics (PK) of CORT118335: Time from Dosing at which Maximum Concentration is Apparent (tmax) | Pre-dose and at pre-specified time points up to 24 hours after dosing on Day 7
Plasma PK of CORT118335: Maximum Observed Concentration (Cmax) | Pre-dose and at pre-specified time points up to 24 hours after dosing on Day 7
Plasma PK of CORT118335: Area Under the Concentration-Time Curve Over the Dose Interval (AUCtau) | Pre-dose and at pre-specified time points up to 24 hours after dosing on Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No